CLINICAL TRIAL: NCT04035915
Title: Comparison Between Limited Driving Pressure Ventilation and Conventional Mechanical Ventilation Strategies in Medical Intensive Care Patients With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI828/2016
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: on Invasive Mechanical Ventilation; ARDS; Respiratory Failure
Keywords: Limited driving pressure; Low tidal volume; Lung injury score
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited driving pressure ventilation (Experimental)
  Interventions: Procedure: Limited driving pressure
- Conventional mechanical ventilation strategies (Experimental)
  Interventions: Procedure: Conventional mechanical ventilation strategies

INTERVENTIONS:
Procedure: Limited driving pressure — Keep driving pressure <15 cmH2O
  Arms: Limited driving pressure ventilation
Procedure: Conventional mechanical ventilation strategies — Keep tidalvolume </= 8
  Arms: Conventional mechanical ventilation strategies

SUMMARY:
Background An appropriated mechanical ventilator setting for acute respiratory failure results of ventilator associated lung injury. Limited driving pressure and low tidal volume ventilation strategies show benefits decreasing mortality in acute respiratory distress syndrome, but there are no data in simple acute respiratory failure.

DETAILED DESCRIPTION:
Background An appropriated mechanical ventilator setting for acute respiratory failure results of ventilator associated lung injury. Limited driving pressure and low tidal volume ventilation strategies show benefits decreasing mortality in acute respiratory distress syndrome, but there are no data in simple acute respiratory failure.

To compare lung injury score (LIS, Murray score) after invasive mechanical ventilation 7 days between groups of limited driving pressure ventilation versus low tidal volume ventilation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year old MICU patient
* On Invasive mechanical ventilator less than 24 hr. before randomization

Exclusion Criteria:

* Suspected death within 48 hr. after randomization
* patients with tracheostomy tube
* Pregnancy
* Do not attempt resuscitation order
* Patient with ECMO before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Lung injury score | Day 7 after invasive mechanical ventilation
  Lung injury score (LIS, Murray score)

SECONDARY OUTCOMES:
28 days Mortality | Upto 28 days
  28 days Mortality
New onset of ARDS | Upto 28 days
  New onset of ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol university, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tongyoo S, Viarasilpa T, Deawtrakulchai P, Subpinyo S, Suppasilp C, Permpikul C. Comparison of limited driving pressure ventilation and low tidal volume strategies in adults with acute respiratory failure on mechanical ventilation: a randomized controlled trial. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241249152. doi: 10.1177/17534666241249152. PMID 38726850